CLINICAL TRIAL: NCT00973934
Title: Magnetic Seizure Therapy (MST) for the Treatment of Major Depression
Acronym: MST-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarah Lisanby (Other)
Collaborators: University of Texas (Other); Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Sarah Lisanby, Professor of psychiatry, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4371; 01-069
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic Seizure therapy (MST) (Experimental): Eligible patients will be randomized to receive either a course of thrice weekly MST using either a focal or non focal stimulating coil.
  Interventions: Device: Magstim Theta
- Right Unilateral Electroconvulsive Therapy (Active Comparator)
  Interventions: Device: Thymatron System IV

INTERVENTIONS:
Device: Magstim Theta
  Arms: Magnetic Seizure therapy (MST)
Device: Thymatron System IV
  Arms: Right Unilateral Electroconvulsive Therapy

SUMMARY:
This two-center, between-subject, randomized, double-masked study (n=20) will provide the first evidence for the antidepressant efficacy of Magnetic Seizure Therapy (MST) and contrast the therapeutic properties and side effects of two forms of MST in patients in a major depressive episode (MDE).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive episode, in the context of unipolar or bipolar disorder
* Age 18-75
* Use of effective method of birth control for women of child-bearing capacity
* Willing and capable of providing informed consent
* Convulsive therapy clinically indicated
* Hamilton Rating Scale for Depression (HRSD) ≥18 (24 item)

Exclusion Criteria:

* Current unstable or serious medical condition, or any comorbid medical condition that substantially increases the risks of ECT (such as acute myocardial infarction, space occupying brain lesion or other cause of increased intracranial pressure, unstable aneurysm or vascular malformation, poorly controlled diabetes mellitus, carcinoma, renal failure, hepatic failure)
* Pregnancy
* History of neurological disorder, epilepsy, stroke, brain surgery, metal in the head, or structural brain lesion
* Presence of devices that may be affected by rTMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Breast-feeding
* History of head trauma with loss of consciousness for greater than 5 minutes
* History of schizophrenia, schizoaffective disorder, or rapid cycling bipolar disorder
* Vagus Nerve Stimulator implanted
* History of substance abuse or dependence in past 3 months
* Failure to respond to an adequate course of ECT in the current depressive episode
* History of ECT in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-04; Primary Completion 2006-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD), 24 item | A blinded rater will administer the test at Baseline, every Tuesday and Thursday during the treatment course and at the end of the MST course

SECONDARY OUTCOMES:
Beck Depression Inventory | A blinded rater will administer the test at Baseline, every Tuesday and Thursady during the treatment course and at the end of the MST course
Neuropsychological testings to assess the acute, short term, long term memory effects of the treatments | A blinded rater will administer various neurospychologiocal tests at various timepoints (baseline, within 3 days following the MST course and at 2 months following the MST course. Treatment Effect Battery (TEB) will be administered at each MST session.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke Universtiy Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914